CLINICAL TRIAL: NCT03257397
Title: Theta-burst Transcranial Magnetic Stimulation for the Treatment of Major Depression
Brief Title: TBS in Major Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rupert Lanzenberger (Other)
Responsible Party: Sponsor-Investigator, Rupert Lanzenberger, Assoc.-Prof. PD Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY-NIL-0008
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left iTBS and right cTBS (Experimental): 40 patients will receive intermittent theta-burst stimulation (iTBS) over the left dorsolateral prefrontal cortex (DLPFC) and continuous TBS (cTBS) over the right DLPFC
  Interventions: Device: theta-burst stimulation (TBS) using a MagPro X1000
- left and right iTBS (Active Comparator): 40 patients will receive intermittent theta-burst stimulation (iTBS) over the left and right dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: theta-burst stimulation (TBS) using a MagPro X1000

INTERVENTIONS:
Device: theta-burst stimulation (TBS) using a MagPro X1000 — iTBS over left and cTBS over right dorsolateral prefrontal cortex for a period of three weeks. iTBS: 3-pulse 50 Hz bursts will be given every 200ms (at 5 Hz) in 2-second trains with an inter-train interval of 8 seconds. cTBS: 3-pulse 50 Hz bursts will be given every 200ms (at 5 Hz) in a single 40s train; one session will comprise left iTBS and right cTBS. There will be two sessions daily with 60 min in between sessions
  Other Names: transcranial magnetic stimulation
  Arms: left iTBS and right cTBS
Device: theta-burst stimulation (TBS) using a MagPro X1000 — iTBS over left and right dorsolateral prefrontal cortex for a period of three weeks. iTBS consists of 3-pulse 50 Hz bursts which will be given every 200ms (at 5 Hz) in 2-second trains with an inter-train interval of 8 seconds. One session will comprise left and right iTBS. There will be two sessions daily with 60 min in between sessions
  Other Names: transcranial magnetic stimulation
  Arms: left and right iTBS

SUMMARY:
Background Major depression is associated with morbidity and increased mortality. Along with the psychological strain depression represents a high socioeconomic burden costing Europe more than €113 billion/year. About one third of patients do not respond to appropriate therapy. Theta-burst stimulation (TBS), a form of transcranial magnetic stimulation is an emerging treatment for patients for whom pharmacological treatment is ineffective or not appropriate. Based on two different theories of prefrontal dysfunction two TBS-protocols should have the most antidepressant effects. However, no study so far has compared the two approaches or systematically investigated their differential effects on brain function and on a symptom level.

Objectives of the study The aim of this study is to test two TBS protocols on symptom improvement and associated brain function in patients with treatment resistant depression (TRD): iTBS over bilateral DLPFC and iTBS over left and cTBS over right DLPFC. As stimulation over non-motor regions offers no direct readout, fMRI at baseline and after treatment will be harnessed to quantify an effect on brain activity and functional network metrics.

Study population 80 patients with TRD will be enrolled with 40 patients receiving the one, and 40 patients receiving the other TBS protocol for a treatment period of three weeks.

Study design The study is designed as a longitudinal, randomized and double-blind clinical trial. At baseline and after treatment, patients will undergo psychiatric testing using several symptom scales including the Hamilton Depression Rating Scale (HAMD-17), the Beck Depression Inventory (BDI-II), the Inventory of Depressive Symptomatology (IDS-C) and the State-Trait Anxiety Inventory (STAI). Changes in HAMD-17 scores are defined as primary endpoint. Moreover MRI scans before and after treatment will include structural and functional MRI sequences as well as diffusion weighted imaging (DWI) sequence. Functional connectivity and BOLD responses will serve as primary imaging endpoints. A follow-up visit 2 weeks and a final examination 4 weeks after treatment will elucidate durability of effects.

Relevance and implications of the study By investigating which approach is superior for which symptoms our study will contribute to the development of personalized treatment, the reduction of personal suffering and the reduction of costs and occupational disability.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of a single or recurrent major depression
* Failure of at least two adequate antidepressant treatments
* HAMD-17 total score of ≥ 23 and a Clinical Global Impression Scale (CGI-S) of ≥ 4
* Stable psychopharmacological treatment within 2 weeks prior inclusion
* Age 18-65 years
* Right-handedness (assessed with the Edinburgh Handedness Inventory)

Exclusion Criteria:

* Seizures in medical history
* Medical history of major systemic illness, neurological disorders and previous brain injuries
* Ferromagnetic implants, cardiac pacemaker, deep brain stimulation and other common MRI and TMS exclusion criteria
* Current psychotic symptoms
* Substance abuse or dependence within last 3 months
* Borderline personality disorder (based on DSM-5 criteria)
* Pregnancy
* Active suicidal intent
* Benzodiazepines other than Lorazepam < 2mg/d
* failure to comply with the study protocol or to follow the instructions of the investigating team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
HAMD | <1 month
  Hamilton depression rating scale
BDI-II | <1 month
  Beck Depression Inventory

SECONDARY OUTCOMES:
Regional white matter microstructure using DWI | <1 month
  White matter microstructure will be investigated using diffusion tensor imaging and analyzed using tract-based spatial statistics and tractography
Regional grey matter volume and using MRI | <1 month
  Regional grey matter volume will be investigated using voxel-based morphometry

OTHER OUTCOMES:
Global physical activity | <1 month
  assessed using Clinical Global Impression Scale (CGI-S)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided